CLINICAL TRIAL: NCT03604458
Title: Evaluating the Impact of Health Insurance on Financial Risk Protection for Surgical Care: an Analysis of Ghana' Insurance Scheme at Korlebu Teaching Hospital
Brief Title: Evaluating the Impact of the National Health Insurance Scheme of Ghana on Surgical Care
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); Fogarty International Center of the National Institute of Health (NIH); University of California Global Health Institute - UCGloCal Program (Unknown); Brigham and Womens' Hospital, Center for Surgery and Public Health (Unknown); UC Global Health Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: D43TW009343 (NIH); D43TW009343 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: General Surgery, Costs and Cost Analysis
Keywords: Universal Health Coverage, Surgery in resource limited settings

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ghana, a Low-Middle Income Country (LMIC) situated in the heart of West Africa started a national health insurance scheme in 2003.The scheme was designed to provide a comprehensive benefit package inclusive of surgical care and to protect against the need to pay out of pocket at the point of service. As of 2013, close to 40% of the population of Ghana was actively enrolled and ongoing plans to expand coverage by the government. This study tests the extent to which the national health insurance scheme of Ghana provides financial risk protection against catastrophic payments as a result of access to surgical care.

DETAILED DESCRIPTION:
It is estimated that 11%-33% of the global burden of disease is attribute to surgical conditions. Yet, globally 3.7 billion people face financial catastrophe if surgical care is needed. Ghana, a country of 27 million people has a 14-year experience with a national health insurance scheme (NHIS) that provides coverage for 95% of the health conditions afflicting Ghanaians and includes access to surgical care. Despite much progress in providing Universal Health Coverage through NHIS, prior work shows that up to 18% of insured households make catastrophic health payments for routine care which is largely unaffordable for the poor. Particularly in Ghana where 1 out of 4 individuals live on less than 1.25 dollars per day. More importantly in 2015, the Lancet Commission on Global Surgery called for national surgical plans that provide 100% coverage against catastrophic health expenditures as a result of seeking surgical care.

The premise of Dr. Okoroh's GloCal project is to describe the surgical conditions that are included in the health insurance scheme and to evaluate whether insurance protect surgical patients against catastrophic health payments through a single institutional review at Korle-bu Teaching Hospital. With this work she hopes to develop a set of recommendations to the ministry of health and the national health insurance authority on how to improve health-care financing for surgical care in Ghana.

Early results of our study show that NHIS provides coverage for most common surgical conditions including symptomatic hernia, breast cancer, and appendicitis. 70% of the total cost of surgical care was covered by NHIS, yet 56% of insured individuals made catastrophic payments for surgical care. Surgery is unaffordable as on average insured individuals spent close to 40% of their annual income on surgical care. Particularly the coverage of medicines, supplies, imaging, and other ancillary services are sparse which are necessary to the provision of surgical care. Our recommendations include; NHIS increasing the proportion of the total cost of surgical care covered for the poor and addressing the gaps in coverage of ancillary services. Further work includes understanding how households economically cope with making payments and the contribution of borrowing and other financing mechanisms in reducing the burden of cost. Our new study characterizes the cost of trauma care which is a major source of disability and injury for young adults in Ghana. Efforts are being made to engage policymakers on healthcare reform in Ghana.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the general surgery ward between February 1st and October 1st 2017.

Exclusion Criteria:

* Patients treated on the subspecialty wards
* Individuals less than 18 years of age.
* If unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was conducted in the Korle Bu teaching hospital, which is situated in the southwestern part of Accra, the capital of Ghana. The hospital receives and treats patients referred from other centers all over Ghana and also patients referred from other neighboring West African countries. The population of Accra, which is largely cosmopolitan, has inhabitants who are natives and a large population who have migrated from other parts of the country on account of economic reason as well as educational pursuit. It is also home to a significant population who are nationals of neighboring West African countries and a small proportion of the population being from Europe, Asia and North America. Inhabitants are therefore mostly urban or suburban with a small proportion of rural and slum dwellers. The Department of Surgery at the Korle Bu hospital has four general surgical units and sees a variety of cases in general surgery encompasses colorectal, hepatobilary, and oncology
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Out of Pocket Expenditure for Surgical Care | During the hospitalization or episode of surgical care (respondents are interviewed prior to discharge from the hospital, on average less than two weeks)
  Out of pocket expenditure for surgical care is defined as all of the direct and indirect expenses incurred by an individual seeking surgical care at Korlebu Teaching Hospital during the study time period.

SECONDARY OUTCOMES:
Catastrophic Health Expenditure for Surgical Care | During the hospitalization or episode of surgical care (respondents are interviewed prior to discharge from the hospital, on average less than two weeks)
  Catastrophic Health Expenditure for Surgical Care is defined as out of pocket expenditures which exceed 20% of the individual's income, 10% of the household expenditures, or 40% of net food expenditures

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Okoroh, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Korle-Bu Teaching Hospital, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okoroh J, Sarpong DO, Essoun S, Riviello R, Harris H, Weissman JS. Does insurance protect individuals from catastrophic payments for surgical care? An analysis of Ghana's National Health Insurance Scheme at Korle-Bu teaching Hospital. BMC Health Serv Res. 2020 Jan 17;20(1):45. doi: 10.1186/s12913-020-4887-2. PMID 31952520